CLINICAL TRIAL: NCT07124286
Title: Does Abdominal Bracing Affect the Upper Extremity Performance in Female Adolescent Volleyball Athletes?
Brief Title: Effects of Abdominal Bracing Maneuver on the Upper Extremity Performance in Volleyball Athletes
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, betül kaya, Research Assistant, Ankara Yildirim Beyazıt University
Other Study IDs: 2023-298
Record Dates: First submitted 2025-08-02; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Upper Extremity Injury
Keywords: Core stabilization; Adolescent athletes; Abdominal bracing maneuver; Functional Performance
MeSH Terms: conditions — Arm Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescent volleyball athletes: Athletes between the ages of 12-18 were recruited as this study has only one group.
  Interventions: Other: Abdominal Bracing Training

INTERVENTIONS:
Other: Abdominal Bracing Training — The group underwent an abdominal bracing maneuver training. Following the training, they performed the Closed Kinetic Chain Upper Extremity Stability Test and the Seated Medicine Ball Throw Test in 2 conditions: with abdominal bracing and without abdominal bracing.

SUMMARY:
The goal of this cross-sectional study is to investigate the effects of abdominal bracing, a trunk co-activation maneuver that activates core muscles, on upper extremity performance tests in adolescent female volleyball athletes. The main question it aims to answer is:

-Does performing the abdominal bracing maneuver increase the upper extremity performance in adolescent female volleyball athletes?

DETAILED DESCRIPTION:
This study aims to determine the acute effects of abdominal bracing maneuver on the stability and strength of the upper extremity. Trunk co-activation maneuvers, also known as volitional preemptive abdominal contraction or abdominal stabilization maneuvers, are developed to prevent and treat spinal instability by boosting core muscle activity. Since core muscles are essential for providing proximal stabilization and maximal force during various activities, take part in the energy transfer between the upper and lower extremities, and reduce the load on the joints; performing the maneuver may increase the athlete's performance.

ELIGIBILITY:
Inclusion Criteria:

* Female adolescent athletes between the ages of 12 and 18
* Attending a volleyball-specific training program at least two times a week
* Not having a systemic and/or neurological disorder
* Not having had a surgery related to upper extremity, lower extremity and/or spine
* Not having had an upper extremity injury for the past six months

Exclusion Criteria:

* Not attending a volleyball-specific training program or attending only once a week
* Having a systemic and/or neurological disorder
* Having had a surgery related to upper extremity, lower extremity and/or spine
* Having had an upper extremity injury for the past six months

Ages: 12 Years to 18 Years | Sex: Female
Age Groups: Child, Adult
Study Population: All participants were female adolescent volleyball athletes between 12 and 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2023-03-25 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Closed Kinetic Chain Upper Extremity Stability Test | Day 1
  Participants were asked to perform the test with and without the abdominal bracing maneuver. Stability of the closed kinetic chain was assessed.
Seated Medicine Ball Throw | Day 1
  Participants were asked to perform the test with and without the abdominal bracing maneuver. Open kinetic chain was assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Betül Kaya, RA, Principal Investigator — Ankara Yildirim Beyazıt University; Zeynep Hazar, Prof., Study Director — Gazi University
Locations (1):
- Gazi University, Ankara, Çankaya, Turkey (Türkiye)

REFERENCES:
- [Background] Aboufazeli M, Afshar-Mohajer N. Within-day and between-day reliability of thickness measurements of abdominal muscles using ultrasound during abdominal hollowing and bracing maneuvers. J Bodyw Mov Ther. 2018 Jan;22(1):122-128. doi: 10.1016/j.jbmt.2017.03.006. Epub 2017 Mar 6. PMID 29332735
- [Background] Ahmed S, Saraswat A, Esht V. Correlation of core stability with balance, agility and upper limb power in badminton players: A cross-sectional study. Sport Sciences for Health. 2022; 18(1): 165-169.
- [Background] Akuthota V, Nadler SF. Core strengthening. Arch Phys Med Rehabil. 2004 Mar;85(3 Suppl 1):S86-92. doi: 10.1053/j.apmr.2003.12.005. PMID 15034861
- [Background] Arora C, Singh P, Varghese V. Biomechanics of core musculature on upper extremity performance in basketball players. J Bodyw Mov Ther. 2021 Jul;27:127-133. doi: 10.1016/j.jbmt.2021.02.023. Epub 2021 Mar 5. PMID 34391223
- [Background] Bauer J, Gruber M, Muehlbauer T. Correlations between core muscle strength endurance and upper-extremity performance in adolescent male sub-elite handball players. Front Sports Act Living. 2022 Nov 10;4:1050279. doi: 10.3389/fspor.2022.1050279. eCollection 2022. PMID 36439625
- [Background] Briner WW Jr, Kacmar L. Common injuries in volleyball. Mechanisms of injury, prevention and rehabilitation. Sports Med. 1997 Jul;24(1):65-71. doi: 10.2165/00007256-199724010-00006. PMID 9257411
- [Background] Chattanooga G 2005 Stabilizer™ pressure bio-feedback. Operating instructions. Hixson: Chattanooga Group Inc.
- [Background] Cigercioglu NB, Guney-Deniz H, Unuvar E, Colakoglu F, Baltaci G. Shoulder Range of Motion, Rotator Strength, and Upper-Extremity Functional Performance in Junior Tennis Players. J Sport Rehabil. 2021 Nov 1;30(8):1129-1137. doi: 10.1123/jsr.2021-0038. Epub 2021 Jul 24. PMID 34303312
- [Background] Davies G, Riemann BL, Manske R. CURRENT CONCEPTS OF PLYOMETRIC EXERCISE. Int J Sports Phys Ther. 2015 Nov;10(6):760-86. PMID 26618058
- [Background] de Araujo RC, Nascimento VYS, Torres RJB, Trombini-Souza F, Behm D, Pitangui ACR. Can the Use of Unstable Surfaces and Instruction for Conscious Abdominal Contraction Increase the EMG Activity of the Periscapular Muscles During the Dynamic Push-Up? J Sport Rehabil. 2020 Feb 1;29(2):225-230. doi: 10.1123/jsr.2018-0165. PMID 30676180
- [Background] Decleve P, Van Cant J, De Buck E, Van Doren J, Verkouille J, Cools AM. The Self-Assessment Corner for Shoulder Strength: Reliability, Validity, and Correlations With Upper Extremity Physical Performance Tests. J Athl Train. 2020 Apr;55(4):350-358. doi: 10.4085/1062-6050-471-18. Epub 2020 Feb 13. PMID 32053404
- [Background] de Villarreal ES, Kellis E, Kraemer WJ, Izquierdo M. Determining variables of plyometric training for improving vertical jump height performance: a meta-analysis. J Strength Cond Res. 2009 Mar;23(2):495-506. doi: 10.1519/JSC.0b013e318196b7c6. PMID 19197203
- [Background] Endo Y, Sakamoto M. Correlation of shoulder and elbow injuries with muscle tightness, core stability, and balance by longitudinal measurements in junior high school baseball players. J Phys Ther Sci. 2014 May;26(5):689-93. doi: 10.1589/jpts.26.689. Epub 2014 May 29. PMID 24926133
- [Background] Ferreira LGR, de Oliveira AS, do Carmo ND, Santos Bueno GA, Lemos TV, Matheus JPC, de Souza Junior JR. Reliability and validity of the One Arm Hop Test and Seated Medicine Ball Throw Test in young adults: A cross-sectional study. J Bodyw Mov Ther. 2021 Oct;28:26-33. doi: 10.1016/j.jbmt.2021.07.018. Epub 2021 Aug 8. PMID 34776150
- [Background] Garcia-Jaen M, Cortell-Tormo JM, Hernandez-Sanchez S, Tortosa-Martinez J. Influence of Abdominal Hollowing Maneuver on the Core Musculature Activation during the Prone Plank Exercise. Int J Environ Res Public Health. 2020 Oct 12;17(20):7410. doi: 10.3390/ijerph17207410. PMID 33053717
- [Background] Gilmer GG, Gascon SS, Oliver GD. Classification of lumbopelvic-hip complex instability on kinematics amongst female team handball athletes. J Sci Med Sport. 2018 Aug;21(8):805-810. doi: 10.1016/j.jsams.2017.12.009. Epub 2018 Jan 9. PMID 29366828
- [Background] Grenier SG, McGill SM. Quantification of lumbar stability by using 2 different abdominal activation strategies. Arch Phys Med Rehabil. 2007 Jan;88(1):54-62. doi: 10.1016/j.apmr.2006.10.014. PMID 17207676
- [Background] Grooms DR, Grindstaff TL, Croy T, Hart JM, Saliba SA. Clinimetric analysis of pressure biofeedback and transversus abdominis function in individuals with stabilization classification low back pain. J Orthop Sports Phys Ther. 2013 Mar;43(3):184-93. doi: 10.2519/jospt.2013.4397. Epub 2012 Nov 16. PMID 23160344
- [Background] Haddas R, Hooper T, James CR, Sizer PS. Volitional Spine Stabilization During a Drop Vertical Jump From Different Landing Heights: Implications for Anterior Cruciate Ligament Injury. J Athl Train. 2016 Dec;51(12):1003-1012. doi: 10.4085/1062-6050-51.12.18. Epub 2016 Nov 22. PMID 27874298
- [Background] Haddas R, Sawyer SF, Sizer PS Jr, Brooks T, Chyu MC, James CR. Effects of Volitional Spine Stabilization and Lower Extremity Fatigue on Trunk Control During Landing in Individuals With Recurrent Low Back Pain. J Orthop Sports Phys Ther. 2016 Feb;46(2):71-8. doi: 10.2519/jospt.2016.6048. Epub 2016 Jan 1. PMID 26721228
- [Background] Jha P, Nuhmani S, Kapoor G, Al Muslem WH, Joseph R, Kachanathu SJ, Alsaadi SM. Efficacy of core stability training on upper extremity performance in collegiate athletes. J Musculoskelet Neuronal Interact. 2022 Dec 1;22(4):498-503. PMID 36458387
- [Background] Kibler WB, Press J, Sciascia A. The role of core stability in athletic function. Sports Med. 2006;36(3):189-98. doi: 10.2165/00007256-200636030-00001. PMID 16526831
- [Background] Kisner C, Colby LA 2007 Therapeutic Exercise: Foundations and Techniques (Fifth Edition). FA Davis Company, Philedelphia.
- [Background] Lidor R, Ziv G. Physical and physiological attributes of female volleyball players--a review. J Strength Cond Res. 2010 Jul;24(7):1963-73. doi: 10.1519/JSC.0b013e3181ddf835. PMID 20543736
- [Background] Maeo S, Takahashi T, Takai Y, Kanehisa H. Trunk muscle activities during abdominal bracing: comparison among muscles and exercises. J Sports Sci Med. 2013 Sep 1;12(3):467-74. eCollection 2013. PMID 24149153
- [Background] Matthijs OC, Dedrick GS, James CR, Brismee JM, Hooper TL, McGalliard MK, Sizer PS Jr. Co-contractive activation of the superficial multifidus during volitional preemptive abdominal contraction. PM R. 2014 Jan;6(1):13-21. doi: 10.1016/j.pmrj.2013.08.606. Epub 2013 Sep 13. PMID 24041586
- [Background] McGill S 2010 Core training: Evidence translating to better performance and injury prevention. Strength and Conditioning Journal 32: 33-46.
- [Background] Nuhmani S. Correlation between Core Stability and Upper-Extremity Performance in Male Collegiate Athletes. Medicina (Kaunas). 2022 Jul 23;58(8):982. doi: 10.3390/medicina58080982. PMID 35893097
- [Background] Pawlik D, Dziubek W, Rogowski L, Struzik A, Rokita A. Strength Abilities and Serve Reception Efficiency of Youth Female Volleyball Players. Appl Bionics Biomech. 2022 Jun 1;2022:4328761. doi: 10.1155/2022/4328761. eCollection 2022. PMID 35694275
- [Background] Pontillo M, Silfies S, Butowicz CM, Thigpen C, Sennett B, Ebaugh D. COMPARISON OF CORE STABILITY AND BALANCE IN ATHLETES WITH AND WITHOUT SHOULDER INJURIES. Int J Sports Phys Ther. 2018 Dec;13(6):1015-1023. PMID 30534467
- [Background] Reeser JC, Verhagen E, Briner WW, Askeland TI, Bahr R. Strategies for the prevention of volleyball related injuries. Br J Sports Med. 2006 Jul;40(7):594-600; discussion 599-600. doi: 10.1136/bjsm.2005.018234. PMID 16799111
- [Background] Saeterbakken AH, van den Tillaar R, Seiler S. Effect of core stability training on throwing velocity in female handball players. J Strength Cond Res. 2011 Mar;25(3):712-8. doi: 10.1519/JSC.0b013e3181cc227e. PMID 20581697
- [Background] Scott R, Yang HS, James CR, Sawyer SF, Sizer PS Jr. Volitional Preemptive Abdominal Contraction and Upper Extremity Muscle Latencies During D1 Flexion and Scaption Shoulder Exercises. J Athl Train. 2018 Dec;53(12):1181-1189. doi: 10.4085/1062-6050-255-17. Epub 2018 Dec 13. PMID 30543446
- [Background] Sheppard JM, Gabbett TJ, Stanganelli LC. An analysis of playing positions in elite men's volleyball: considerations for competition demands and physiologic characteristics. J Strength Cond Res. 2009 Sep;23(6):1858-66. doi: 10.1519/JSC.0b013e3181b45c6a. PMID 19675472
- [Background] Shinkle J, Nesser TW, Demchak TJ, McMannus DM. Effect of core strength on the measure of power in the extremities. J Strength Cond Res. 2012 Feb;26(2):373-80. doi: 10.1519/JSC.0b013e31822600e5. PMID 22228111
- [Background] Silva AF, Clemente FM, Lima R, Nikolaidis PT, Rosemann T, Knechtle B. The Effect of Plyometric Training in Volleyball Players: A Systematic Review. Int J Environ Res Public Health. 2019 Aug 17;16(16):2960. doi: 10.3390/ijerph16162960. PMID 31426481
- [Background] Swanik KA, Lephart SM, Swanik CB, Lephart SP, Stone DA, Fu FH. The effects of shoulder plyometric training on proprioception and selected muscle performance characteristics. J Shoulder Elbow Surg. 2002 Nov-Dec;11(6):579-86. doi: 10.1067/mse.2002.127303. PMID 12469083
- [Background] Tucci HT, Martins J, Sposito Gde C, Camarini PM, de Oliveira AS. Closed Kinetic Chain Upper Extremity Stability test (CKCUES test): a reliability study in persons with and without shoulder impingement syndrome. BMC Musculoskelet Disord. 2014 Jan 3;15:1. doi: 10.1186/1471-2474-15-1. PMID 24387196
- [Background] Vega Toro AS, Cools AM, de Oliveira AS. Instruction and feedback for conscious contraction of the abdominal muscles increases the scapular muscles activation during shoulder exercises. Man Ther. 2016 Sep;25:11-8. doi: 10.1016/j.math.2016.05.331. Epub 2016 Jun 1. PMID 27422592
- [Background] Vera-Garcia FJ, Elvira JL, Brown SH, McGill SM. Effects of abdominal stabilization maneuvers on the control of spine motion and stability against sudden trunk perturbations. J Electromyogr Kinesiol. 2007 Oct;17(5):556-67. doi: 10.1016/j.jelekin.2006.07.004. Epub 2006 Sep 22. PMID 16996278
- [Background] Warren L, Baker R, Nasypany A, Seegmiller J 2014 Core concepts: understanding the complexity of the spinal stabilizing systems in local and global injury prevention and treatment. International Journal of Athletic Therapy and Training 19: 28-33.
- [Background] Weston M, Hibbs AE, Thompson KG, Spears IR. Isolated core training improves sprint performance in national-level junior swimmers. Int J Sports Physiol Perform. 2015 Mar;10(2):204-10. doi: 10.1123/ijspp.2013-0488. Epub 2014 Jul 8. PMID 25025936